CLINICAL TRIAL: NCT05910632
Title: Effect of Eight Weeks of Eccentrically Reinforced Resistance Training Versus Traditional Resistance Training on Depressive Symptoms, Physical and Executive Function in Sedentary Older Women
Brief Title: Eccentrically Reinforced Resistance Training vs. Traditional Resistance Training in Sedentary Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Vicosa (Other)
Responsible Party: Principal Investigator, Édison Andrés Pérez Bedoya, Principal Investigator, Federal University of Vicosa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Resistance exercise - UFV
Record Dates: First submitted 2023-05-15; First posted 2023-06-20 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Depression; Physical Functional Performance; Executive Function
Keywords: Depression; Physical Function; Executive Function
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Hidden and opaque envelope technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentrically strengthened resistance exercise (Experimental): Women who will be part of the eccentrically reinforced resistance group will perform using the multi-gym equipment with flywheel. Each workout will involve upper and lower extremities.
  Interventions: Behavioral: Eccentrically strengthened resistance exercise
- Traditional resistance training (Active Comparator): The control group (traditional resistance program) will carry out their interventions on gym machines for the lower limbs and free weights for the upper extremities.
  Interventions: Behavioral: Traditional resistance training

INTERVENTIONS:
Behavioral: Eccentrically strengthened resistance exercise — For each resistance exercise session, 6 to 7 generic exercises will be performed, involving small and large muscle groups (leg extension, leg curl, biceps curl, triceps extension, seated row, shoulder flexion, and shoulder raise). They will perform with 4 sets of 8 repetitions, with a break between exercises of 1 minute and between sets of 2 minutes. They perform those exercises with high intensity (ever 10 on the OMNI-RES Scale).
  Arms: Eccentrically strengthened resistance exercise
Behavioral: Traditional resistance training — For each resistance exercise session, 6 to 7 generic exercises will be performed, involving small and large muscle groups (leg extension, leg curl, biceps curl, triceps extension, seated row, shoulder flexion, and shoulder raise). They will perform with 4 sets of 8-12 repetitions, with a break between exercises of 1 minute and between sets of 2 minutes. They perform those exercises with moderate and high intensities (6 to 10 on the OMNI-RES scale).
  Arms: Traditional resistance training

SUMMARY:
There are easily accessible and safe strategies, such as physical exercise, that can contribute to reducing depressive symptoms and to the preservation of physical and executive function in elderly women. Resistance exercise is defined as performing in water or on land. It involves exercise using a constant load or a uniform weight regardless of the training program. There are many types of resistance exercise equipment, including free weights, pneumatic resistance machines, and elastic bands. Specifically, eccentric muscle contraction occurs when the force applied to the muscle exceeds the momentary force produced by the muscle itself, resulting in forced lengthening of the muscle-tendon system while contracting.

To date, a body of evidence has been found derived from randomized controlled trials, which have compared the effectiveness of aerobic, resistance exercise and Pilates in decreasing depressive symptoms and improving physical and executive function in elderly women.

Although there are experimental studies demonstrating the effectiveness of physical exercise, the effect of short-term eccentrically reinforced strength training on depressive symptoms, physical and executive function in sedentary older women is unclear.

Therefore, this study aims to evaluate the safety and effect of eccentrically reinforced resistance exercise vs. traditional resistance training on depressive symptoms, physical and executive function, quality of life, different manifestations of muscle strength, body composition, vital signs and abdominal circumference, risk of falls, quality of sleep sedentary older women for 8 weeks.

DETAILED DESCRIPTION:
Twenty-two women will be randomly assigned to two groups (eccentrically enhanced resistance training and traditional resistance training). Interventions will be conducted in the Department of physical education of federal university of Viçosa. All sessions will be supervised by physical education professors. Follow-up will be done through WhatsApp messages and phone calls. Both groups will have a training frequency of 2 times per week for eight weeks. Eccentrically augmented resistance sessions will be performed on the multi-gym flywheel machine for lower and upper limbs for women in the experimental group. The control group will use machines and free weights. In each training session, 6 to 7 exercises will be performed, with 4 sets of 8-12 repetitions, with a rest between exercises of 1 minute and between sets of 2 minutes. The resistance exercise progression is carried out until the woman, with the same mobilized weight in kg, exceeds the maximum number of repetitions suggested by the researchers. Each resistance exercise session will include 6-7 generic exercises involving small and large muscle groups (leg extension, leg curl, biceps curl, triceps extension, seated row, shoulder flexion, and shoulder raise).

Each participant will undergo an initial and final assessment to measure the muscle strength of the lower extremities. The depressive state will be evaluated with a short version of the Geriatric Depression Scale (GDS), validated in Brazil. The physical function will be evaluated with the Test Timed Up and Go (TUG) and Short Physical Performance Battery (SPPB). In addition, executive function will be evaluated with the Victoria Stroop test. Work memory, Digit span forward, Backward and Cognitive flexibility with Trail marking test (Trail A and Trail B).

The Brazilian version of WHOQOL-Bref will be used to assess quality of life. To evaluate the maximum isometric voluntary contraction (MIVC) of the lower extremities, a load cell or extensiometric cell (MK®, model CSL / ZL-1 T, MK Controle, Brazil) with a sampling frequency of 1000 Hz will be used. To perform the 1RM test, the knee extension exercise is performed on a BH fitness® Nevada Pro-t extension machine. The evaluation of lower limb muscular strength will be performed with the same knee extension machine used in training sessions, starting from the same initial position (90o knee flexion) and reaching. Body composition is assessed using a dual-energy x-ray absorptiometry (DXA) full-body scan (GE Healthcare Lunar Prodigy Advance DXA System, software version 13.31). A minimus® III aneroid sphygmomanometer with a maximum error of +/- 3 mmHg will be used. Systolic blood pressure (SBP), diastolic blood pressure (DBP), and mean blood pressure (MBP) are calculated. MBP is obtained with the following mathematical operation: PAD + PAD + PAS / 3. To measure HRR, women are asked to sit for 3 minutes. After that moment, this variable will be taken manually in the radial or carotid pulse of the right side for 60 seconds. The perimeter of the abdomen is measured with a metal tape with the subject's feet, at a midpoint between the lower costal margin and the iliac crest, at the end of a normal expiration.

The risk of falling will be evaluated with the Falls Efficacy Scale-International (FES-I).

Sleep-wake cycle evaluation with Actigraph GT3X-BT Accelerometer Sleep Quality Assessment: Pittsburg Sleep Quality Index - PSQI Chronotype Assessment: Hortensia and Ostberg Questionnaire Sleepiness Assessment: Epworth Sleepiness Scale.

ELIGIBILITY:
Inclusion Criteria:

1. 60 years or older.
2. Self-reported proficiency in speaking, writing, and understanding Portuguese.
3. Willingness and availability to participate in all trial procedures.
4. Good vision in at least one eye.
5. Absence of any medical contraindications for engaging in physical exercise.
6. Engage in less than 150 minutes of physical activity per week.
7. Not clinical diagnosis of major depressive disorder at the time of the interventions.

Exclusion Criteria:

1. Elderly women with uncontrolled chronic diseases.
2. Clinical diagnosis of psychiatric illness.
3. Women who have undergone or are expected to undergo surgical procedures during the interventions.
4. Elderly women diagnosed with joint diseases such as osteoarthritis and arthrosis.
5. Participation in aerobic or resistance exercise programs at least 2 times a week for the past 3 months.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in baseline depressive symptoms at two months. | Baseline and 8-weeks
  Test: The depressive state will be evaluated with a short version of the validated geriatric depression scale (GDS) in Brazil. There are 15 questions that inquire about feelings and a frequency that the person presents before certain conditions of life. These questions require categorical answers (yes or no). Of the 15 items, 10 indicate the presence of depression when answered positively. While the rest (1, 5, 7, 11 and 13) when answered negatively. A higher score indicates depression.
Change in baseline test Time up and go at two months. | Baseline and 8-weeks
  Test: The time up and go will assess sitting balance, balance in transfers from sitting to standing, stability in ambulation and changes of direction. The test consists of the individual getting up from the chair, without arm support, walking 3 meters with safe and comfortable steps, without running, turning 180°, returning and sitting in the chair. The time taken to perform this task will be timed. Volunteers who perform the task in a time of less than 10 seconds will be considered with satisfactory mobility, for those who perform the test between 11 and 20 seconds will be classified with good mobility and for those who reach values greater than 20 seconds will be classified with mobility problems.
Change in baseline balance test, mark speed, and sit and stand chair at two months | Baseline and 8-weeks
  The Short Physical Performance Battery (SPPB) in its Brazilian version will be performed, which includes the tests for standing static balance, gait speed, and lower limb muscle strength. The total score of the SPPB will be obtained by adding the score of each test, ranging from zero (worst capacity) to 12 (best capacity). The result can be graded as follows: 0 to 3 points: disability or poor capacity; 4 to 6 points: low capacity; 7 to 9 points: moderate capacity; and 10 to 12 points: good capacity.
Change in Inhibitory control at two months | Baseline and 8-weeks
  Test: Victoria Stroop test. Inhibitory control will be evaluated using the Victoria Stroop Test, which uses three tasks with 24 items each. The participant is evaluated according to how quickly she performs the task and the number of errors. The effect of interference is determined by calculating the extra time required to name the colors (of the printout) compared to the time required to name colors in the first control task (colors of the cards). The task performed faster indicates better performance.
Change in Working memory at two months | Baseline and 8-weeks
  Working memory will be evaluated by Digit Span Forward and Backward. For the calculation of the test, the sum of the longest sequence of digits repeated, without error, over two trials in direct order is used.
Change in Cognitive flexibility at two months | Baseline and 8-weeks
  Test composed of two parts (Tracks A and Tracks B). The execution time for each of the tests is limited to four minutes or three errors The test score will be obtained through the time spent to finish each part. For speed adjustment, the difference between the completion times of part B and part A will be calculated, in which smaller differences in scores indicate better speed adjustments.

SECONDARY OUTCOMES:
Change in baseline quality of life time at two months. | Baseline and 8-weeks
  Test: World Health Organization Quality of Life Assessment Bref. The Brazilian version of the World Health Organization Quality of Life Assessment Bref will be utilized in this study. The 26 items produce 4 domains related to Quality of Life; physical (health), psychological, social relationships and environmental and an overall Quality of life and health satisfaction facet. Each item is measured from 1 to 5 on a Likert scale, with varying scale response anchors, where higher values represent higher Quality of life. One example of item is "How much do you enjoy life?", rated on the following response options (1) not at all, (2) a little, (3) a moderate amount, (4) very much, and (5) an extreme amount.
Maximum isometric voluntary contraction | Baseline and 8-weeks
  To evaluate the Maximum isometric voluntary contraction (MIVC) of the lower extremities, a load cell or extensiometric cell (MK®, CSL / ZL-1 T, MK Controle, Brazil) with a sampling frequency of 1000 Hz will be used.
1RM test | Baseline and 8-weeks
  To perform the one repetition maximum test (1RM), the knee extension exercise will be used on a BH fitness® Nevada Pro-t extension machine. To perform the test, the volunteer will be asked to extend the knee to form an angle of approximately 180° (final position) and return to the initial position.
Muscle power | Baseline and 8-weeks
  The evaluation of lower limb muscle power will be performed using the same knee extension machine used in the exercise sessions, starting from the same initial position (90º of kneeling flexion) and reaching the same final position (180º of knee extension) as the test of 1RM.
Change In Baseline Total body mass at two months | Baseline and 8-weeks
  Dual-engy X-ray absorptiometry (DXA) full body exam (GE Healthcare Lunar Prodigy Advance DXA System, software version 13.31).
Change In Baseline lean mass At Two Months | Baseline and 8-weeks
  Dual-engy X-ray absorptiometry (DXA) full body exam (GE Healthcare Lunar Prodigy Advance DXA System, software version 13.31).
Change In Baseline bone mineral content At Two Months | Baseline and 8-weeks
  Dual-engy X-ray absorptiometry (DXA) full body exam (GE Healthcare Lunar Prodigy Advance DXA System, software version 13.31).
Change In Baseline bone mineral density At Two Months | Baseline and 8-weeks
  Dual-engy X-ray absorptiometry (DXA) full body exam (GE Healthcare Lunar Prodigy Advance DXA System, software version 13.31).
Change In Baseline bone loss index throughout life At Two Months | Baseline and 8-weeks
  Dual-engy X-ray absorptiometry (DXA) full body exam (GE Healthcare Lunar Prodigy Advance DXA System, software version 13.31).
Blood pressure | Baseline and 8-weeks
  minimus® III aneroid tensiometer will be used, which has a maximum error margin of +/-3 mmHg. Systolic blood pressure (SBP), diastolic blood pressure (DBP), and mean blood pressure (MBP) will be calculated. MBP will be obtained with the following mathematical operation: PAD + PAD + PAS / 3
Resting heart rate | Baseline and 8-weeks
  For Resting heart rate (HRR) measurement, women will be advised to sit for 3 minutes. After that moment, this variable will be taken manually in the radial or carotid pulse of the right side for 60 seconds.
Abdominal circumference | Baseline and 8-weeks
  Metallic tape measure
Number of participants with adverse events or damages | 8-weeks
  A self-designed questionnaire consisting of categorical questions (yes or no) will be utilized to assess adverse events. The severity of adverse events will be graded using version 5.0 of the "Common Terminology Criteria for Adverse Events" (CTCAEv5.0). Possible adverse events related to the intervention will be documented in the questionnaire.
Change in baseline Falls Efficacy Scale-International at to months | Baseline and 8-weeks
  The risk of falling will be assessed by means of the Falls Efficacy Scale-International (FES-I) questionnaire in its Brazilian version, which evaluates the concern with the possibility of falling when performing 16 activities, with respective scores from one to four. The total score can vary from 16 (no concern) to 64 (extreme concern).
Changes in baseline active time at two months. | Baseline and 8-weeks
  For the actimetry the Actigraph GT3X-BT accelerometer will be used for a period of eight days. The participant must fill out a sleep diary together with the use of the accelerometer. The ActiLive software will be used to analyze active time (minutes). The sleep diary will be used for possible adjustments in the quantification of the reading variables. The results of the analysis will allow the identification of sleep time and its quality, according to the time of latency and awakenings throughout the night, and whether the participant can maintain a sleep-wake pattern.
Changes In Baseline Sleep latency At Two Months. | Baseline and 8-weeks
  For the actimetry the Actigraph GT3X-BT accelerometer will be used for a period of eight days. The participant must fill out a sleep diary together with the use of the accelerometer. The ActiLive software will be used to analyze sleep latency (minutes) The sleep diary will be used for possible adjustments in the quantification of the reading variables. The results of the analysis will allow the identification of sleep time and its quality, according to the time of latency and awakenings throughout the night, and whether the participant can maintain a sleep-wake pattern.
Changes in baseline sleep quality at two months. | Baseline and 8-weeks
  The Pittsburg Sleep Quality Index will be used to evaluate the subjective quality of sleep and the presence of sleep disturbances in a period of four weeks prior to its application. In relation to the score, when the score is less than 5 it indicates the absence of sleep disturbances or a good quality of sleep, and when the sum is greater than 5 points it indicates a poor quality of sleep and possible presence of sleep disturbances. A sum closer to 0 indicates better quality and no sleep disturbance.
Changes In Baseline Wakefulness after sleep onset At Two Months. | Baseline and 8-weeks
  For the actimetry the Actigraph GT3X-BT accelerometer will be used for a period of eight days. The participant must fill out a sleep diary together with the use of the accelerometer. The ActiLive software will be used to analyze wakefulness after sleep onset (minutes). The sleep diary will be used for possible adjustments in the quantification of the reading variables. The results of the analysis will allow the identification of sleep time and its quality, according to the time of latency and awakenings throughout the night, and whether the participant can maintain a sleep-wake pattern.
Changes in baseline chronotype at two months. | Baseline and 8-weeks
  Changes in chronotype at baseline and in eight weeks. For the analysis of the chronotype profile, the Horne and Ostberg questionnaire will be used, consisting of 19 questions. It will classify the participants into afternoon, intermediate, and morning. Scores can range from 16-86. Scores of 41 and below indicate "afternoon types"; scores of 59 and above indicate "morning types," and scores between 42-58 indicate "intermediate types."
Changes In Baseline Total sleep time At Two Months. | Baseline and 8-weeks
  For the actimetry the Actigraph GT3X-BT accelerometer will be used for a period of eight days. The participant must fill out a sleep diary together with the use of the accelerometer. The ActiLive software will be used to analyze total sleep time (minutes) The sleep diary will be used for possible adjustments in the quantification of the reading variables. The results of the analysis will allow the identification of sleep time and its quality, according to the time of latency and awakenings throughout the night, and whether the participant can maintain a sleep-wake pattern.
Changes In Baseline Sleep efficiency At Two Months. | Baseline and 8-weeks
  For the actimetry the Actigraph GT3X-BT accelerometer will be used for a period of eight days. The participant must fill out a sleep diary together with the use of the accelerometer. The ActiLive software will be used to analyze sleep efficiency (%). The sleep diary will be used for possible adjustments in the quantification of the reading variables. The results of the analysis will allow the identification of sleep time and its quality, according to the time of latency and awakenings throughout the night, and whether the participant can maintain a sleep-wake pattern.
Changes in baseline sleepiness at two months | Baseline and 8-weeks
  The Epworth Sleepiness Scale subjectively assesses an individual's levels of sleepiness. Higher scores indicate abnormal sleepiness. Scores: 1-6 points (Normal sleep); 7-8 points (Average sleepiness) and 9-24 points (Abnormal sleepiness).

CONTACTS AND LOCATIONS:
Overall Officials: Édison A. Pérez Bedoya, PhD, Principal Investigator — Federal University of Vicosa
Locations (1):
- Federal University of Viçosa, Viçosa, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andres Perez Bedoya E, Puerta-Lopez LF, Garcia Agostinho PA, Reis Cota AD, Patrocinio de Oliveira CE, Araujo Carneiro-Junior M, Patino-Villada FA, Costa Moreira O. Flywheel resistance training and depressive symptoms in older women: a randomized controlled trial. Aging Ment Health. 2025 Nov 7:1-14. doi: 10.1080/13607863.2025.2575025. Online ahead of print. PMID 41202328